CLINICAL TRIAL: NCT03601754
Title: Effectiveness of Closed Loop Stimulation (CLS) With His Bundle Lead Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-00143
Record Dates: First submitted 2018-05-02; First posted 2018-07-26 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Sinus Node Dysfunction
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Closed Loop Stimulation (CLS) (Experimental): Prior to enrollment, the patient would have received Biotronik pacemaker with His bundle lead placement for at least 30 days and CLS will be programmed ON for at least 7 days as part of routine care.
  Interventions: Diagnostic Test: Treadmill/Bicycle exercise testing

INTERVENTIONS:
Diagnostic Test: Treadmill/Bicycle exercise testing — Exercise testing will be scheduled on the same day as the enrollment visit and within 30 days after post-implant visit.
  The standard protocol will be typically set at an initial workload of 15Watts and go up by increments of 10 Watts every 3 minutes, as follows:
  Stage 1 - 15 W Stage 2 - 25 W Stage 3 - 35 W Stage 4 - 45 W

SUMMARY:
This study is a prospective, non-randomized pilot study looking to evaluate the effectiveness of Closed Loop Stimulation (CLS) in sinus node dysfunction patients with HIS bundle placement. Patients with sinus node dysfunction who have previously received a Biotronik pacemaker with His bundle lead placement as part of routine care will be recruited for the study. A hand-grip exercise will be performed at the conclusion of bicycle exercise testing in order to assess the performance of CLS during isometric exercise. After the study exercise testing is completed, data will be collected from the pacemaker.

ELIGIBILITY:
Inclusion Criteria:

* Documented sinus node dysfunction
* Biotronik pacemaker implanted with His bundle lead placement for standard indications
* Implanted at least 30 days
* CLS has been enabled for at least 7 days or will be programmed ON for at least 7 days prior to exercise test
* Leads and device are functioning appropriately

Exclusion Criteria:

* Inability to complete treadmill/bicycle exercise test
* Planned surgical revision or replacement of the device and/or leads
* Patients who are unwilling or unable to provide informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Change in heart rate from baseline to Day 30 | Day 1, Day 30
  Ability to achieve adequate heart rate, defined as reaching upper sensor rate, during peak exertion

SECONDARY OUTCOMES:
Greater heart response with CLS compared to predicted accelerometer based heart rate response | Day 1, Day 30
  CLS rate response will be analyzed individually for each subject by comparing the CLS response, which is collected by the CLS Action Log, to heart rate information.

CONTACTS AND LOCATIONS:
Overall Officials: Chirag Barbhaiya, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States